CLINICAL TRIAL: NCT05431413
Title: Fluoxetine Combined With ATP Rapidly Improves Moderate to Severe Depression: a Pilot Study
Brief Title: Rapid Improvement of Depression of Fluoxetine Combined With ATP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2020-153
Record Dates: First submitted 2022-06-12; First posted 2022-06-24 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Adenosine Triphosphate; Phosphocreatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group: Fluoxetine and Placebo (Placebo Comparator): Cap Fluoxetin 20mg OD for four weeks and injection 100ml normal saline(NS) BD for two weeks.
  Interventions: Drug: Control group: Fluoxetine and Placebo
- Experimental group: Fluoxetine and ATP (Experimental): Cap Fluoxetin 20mg OD for four weeks and injection ATP 100mg in NS BD for two weeks.
  Interventions: Drug: Experimental group: Fluoxetine and ATP
- Control group: Fluoxetine and Phosphocreatine (Active Comparator): Cap Fluoxetin 20mg OD for four weeks and injection phosphocreatine(1g) in NS BD for two weeks.
  Interventions: Drug: Control group: Fluoxetine and Phosphocreatine

INTERVENTIONS:
Drug: Control group: Fluoxetine and Placebo — Cap Fluoxetin 20mg OD for four weeks and injection 100ml normal saline(NS) BD for two weeks.
  Arms: Control group: Fluoxetine and Placebo
Drug: Experimental group: Fluoxetine and ATP — Cap Fluoxetin 20mg OD for four weeks and injection ATP 100mg in NS BD for two weeks.
  Arms: Experimental group: Fluoxetine and ATP
Drug: Control group: Fluoxetine and Phosphocreatine — Cap Fluoxetin 20mg OD for four weeks and injection Phosphocreatine 1g in NS BD for two weeks.
  Arms: Control group: Fluoxetine and Phosphocreatine

SUMMARY:
The clinical study is a randomized (1:1:1), double-blind, placebo-controlled clinical study. Recruit patients with moderate to severe depression. After signing the informed consent, patients who meet the inclusion criteria will be randomly assigned to the ATP group (fluoxetine combined with ATP) or phosphocreatine group (fluoxetine combined with phosphocreatine) or control group (fluoxetine combined with 0.9% sodium chloride) to received treatment. Then accessed scale, cognitive function and brain function before treatment and at one, two, and four weeks after treatment to initially explore the safety and efficacy of ATP combined with fluoxetine to rapidly improves moderate to severe depression.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-V diagnostic criteria for moderate to severe depression.
* HAMD-24 scores ≥ 20.
* 18-65 female or male.
* Subjects who have not used any antipsychotic drugs, antidepressants, mood stabilizers (sodium valproate, lithium carbonate) or fluoxetine treatment within the first month prior to the start of this study
* Written informed consent.

Exclusion Criteria:

* Sufferring from various major mental disorders other than depression (such as bipolar disorder, schizophrenia, personality split, etc.).
* Individuals with neurological disorders such as dementia.
* Individuals with a high risk of suicide.
* Pregnant and lactating women.
* Individuals with alcohol or drug abuse or dependence within one year prior to the start of this study.
* Contraindications to MRI.
* Physician evaluation was not suitable for participants in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale | Baseline and one, two, four weeks after treatment
  Changes in Hamilton Depression Scale（HAMD-24）

SECONDARY OUTCOMES:
structural brain networks | Baseline and two, four weeks after treatment
  Changes in diffusion tensor imaging（DTI）and Diffusion Spectral Imaging(DSI)
functional brain networks | Baseline and two and four weeks after treatment
  Changes in functional magnetic resonance imaging（fMRI）and quantitative susceptibility mapping(QSM）
Hamilton Anxiety Scale | Baseline and one, two, four weeks after treatment
  Changes in Hamilton Anxiety Scale（HAMA）
Clinical Global Impression | Baseline and one, two, four weeks after treatment
  Changes in Clinical Global Impression（CGI）
Snaith-Hamilton Pleasure Scale | Baseline and one, two, four weeks after treatment
  Changes in Snaith-Hamilton Pleasure Scale（SHAPS）
Insomnia Severity Index | Baseline and one, two, four weeks after treatment
  Changes in Insomnia Severity Index（ISI）
Patient Health Questionnaire | Baseline and one, two, four weeks after treatment
  Changes in Patient Health Questionnaire（PHQ-9）
Columbia-Suicide Severity Rating Scale | Baseline and one, two, four weeks after treatment
  Changes in Columbia-Suicide Severity Rating Scale（C-SSRS)
Antidepressants Side Effects | Baseline and one, two, four weeks after treatment
  Number of Participants with antidepressants side effects（SERS）
C-reaction protein | Baseline and two and four weeks after treatment
  Changes in C-reaction protein（CRP）
Tumor Necrosis Factor α | Baseline and two and four weeks after treatment
  Changes in Tumor Necrosis Factor（TNF-α）
interleukin- 6 | Baseline and two and four weeks after treatment
  Changes in interleukin- 6（IL-6）
N-back task | Baseline and two and four weeks after treatment
  Changes in reaction time and accuracy
Stroop task | Baseline and two and four weeks after treatment
  Changes in reaction time and accuracy
Psychomotor vigilance task | Baseline and two and four weeks after treatment
  Changes in reaction time and accuracy
Attention network test | Baseline and two and four weeks after treatment
  Changes in reaction time and accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zhang, MD & PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China